CLINICAL TRIAL: NCT06859593
Title: Comparison Of Upper Extremity Exercise Capacity Of Breast Cancer Patients With Healthy Individuals
Brief Title: Upper Extremity Exercise Capacity Of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Professor, Hacettepe University
Other Study IDs: FTREK 25/01
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Survivor; Healty Controls
Keywords: breast cancer; upper extremity; 6-minute pegboard and ring test; exercise capacity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast Cancer Group: Inclusion criteria were to be between 18-65 years of age, to volunteer to participate in the study, to have Stage I-III breast cancer, to have at least 15 months after breast cancer surgery, to have six months after active breast cancer treatment (i.e. surgery/chemotherapy), to have no problems in reading and/or understanding the scales and to be able to cooperate with the tests. Exclusion criteria were the presence of active infection, musculoskeletal and neurologic disease that may affect exercise performance, symptomatic heart disease, neurologic disease or other clinical diagnosis that may affect cognitive status.
  Interventions: Diagnostic Test: Upper Extremity Exercise Capacity, 6-Minute Pegboard And Ring Test
- Control Group: The inclusion criteria were to be between 18-65 years of age, to be willing to participate in the study, to have no problems in reading and/or understanding the scales and to be able to cooperate with the tests. Exclusion criteria were having any orthopedic or neuromuscular condition that would interfere with walking or exercise performance, having any chronic disease, or having psychiatric disorders or mental disorders that might interfere with cooperation or compliance with exercise tests.
  Interventions: Diagnostic Test: Upper Extremity Exercise Capacity, 6-Minute Pegboard And Ring Test

INTERVENTIONS:
Diagnostic Test: Upper Extremity Exercise Capacity, 6-Minute Pegboard And Ring Test — Upper Extremity Exercise Capacity

SUMMARY:
Breast cancer is one of the most common cancers among women worldwide, with an incidence rate of up to 16%. Although survival can be improved with early diagnosis and more effective therapies, physical complications such as lymphedema, upper extremity dysfunction and chronic pain are common during and/or after breast cancer treatments. In addition, lymphedema can cause symptoms such as decreased muscle strength and range of motion of the upper extremity, pain and fatigue, resulting in activity limitations and decreased functional level of the upper extremity.

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers among women worldwide, with an incidence rate of up to 16%. While the breast cancer survival rate is 80% in developed countries, this rate varies between 40-60% in low-middle income countries. Although survival can be increased with early diagnosis and more effective therapies, physical complications such as lymphedema, upper extremity dysfunction and chronic pain are frequently observed during and/or after breast cancer treatments. Upper extremity lymphedema that develops after breast cancer treatment usually affects the glenohumeral joint by increasing the tension in the tendons of the rotator cuff muscles and disrupting the scapulohumeral rhythm. In addition, lymphedema may cause symptoms such as decreased muscle strength and range of motion of the upper extremity, pain and fatigue, resulting in activity limitations and decreased functional level of the upper extremity. Kinesiophobia (fear-avoidance reaction to activity), which may develop in patients in relation to the affected extremity, is another factor in decreased capacity of the upper extremity. Patients may restrict the use of their extremities to prevent aggravation of lymphedema. Decreased functional capacity is common after breast cancer treatment. The '6 Minute Pegboard and Ring Test-6PBRT' is a valid and reliable, useful, practical and easy-to-administer test that evaluates unsupported arm endurance in breast cancer patients, patients with COPD, patients with asthma and healthy individuals. For the test, patients are asked to carry as many rings as possible within 6 minutes and the number of rings carried for 6 minutes is recorded as a score. In a study conducted in patients with mild to very severe COPD, it was shown that there was a positive correlation between the 6PBRT score and activity counts assessed by accelerometry. In addition, the 6PBRT score showed a clear relationship with upper extremity ROM and it was concluded that the 6PBRT test can be used as a suitable test for predicting and demonstrating improvement of ROM in pulmonary rehabilitation programs. Therefore, the aim of this study was to test both arm endurance and arm exercise capacity of patients with breast cancer using the 6PBRT test and to compare them with healthy individuals to understand how much they are affected compared to healthy individuals.

As a secondary aim of the study, it is planned to investigate the relationship between lymph edema severity and anthropometric measurements and upper extremity activities and arm exercise capacity in the group with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Breast Cancer Group:

1. Being between 18-65 years of age,
2. Volunteering to participate in the research,
3. Stage I-III breast cancer,
4. At least 15 months after breast cancer surgery,
5. Six months after active breast cancer treatment (i.e. surgery/chemotherapy),
6. No problems in reading and/or understanding the scales and being able to cooperate with the tests,

Healthy group:

1. Age between 18-65 years,
2. Volunteering to participate in the research,
3. No problems in reading and/or understanding the scales and being able to cooperate with the tests.

Exclusion Criteria:

Breast Cancer Group:

1. Presence of active infection,
2. Musculoskeletal and neurological diseases that may affect exercise performance, symptomatic heart disease,
3. Having a neurological disease or other clinical diagnosis that may affect cognitive status.

Healthy group:

1. Having any orthopedic or neuromuscular condition that would interfere with walking or exercise performance,
2. Having any chronic disease or psychiatric disorders or mental impairments that may interfere with cooperation or compliance with exercise tests

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 years who are diagnosed with breast cancer at Hacettepe University Hospital, Department of Internal Medicine, Division of Medical Oncology, and who volunteer to participate in the study will be included in the study. For healthy groups, age and gender appropriate volunteers will be recruited for the study
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Exercise Capacity | One Year
  6-Minute Pegboard and Ring Test

SECONDARY OUTCOMES:
Evaluation of Upper Extremity Functionality | One Year
  Questionnaire Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) The score ranges from 0 to 100. A higher score reflects more severe upper extremity dysfunction, and the cutoff scores are 0-15 for normal, 16-40 for having problems but working, and more than 40 for being unable to work
Lymphedema Evaluation | One Year
  Arm circumference measurement
Measurement of arm length, arm and forearm circumference | One Year
  The circumference and length measurements of the participants' dominant and non-dominant arm will be measured using a tape measure

CONTACTS AND LOCATIONS:
Overall Officials: Melda Saglam, PhD, Study Chair — Hacettepe University
Locations (1):
- Hcettepe University, Ankara, State 06100, Ankara, State, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No